CLINICAL TRIAL: NCT04589585
Title: Merlin's DiVeRt-Vascular Reconstruction Device: a Prospective, Single Arm, Non-randomized, Open Label Study to Assess Safety and Performance
Brief Title: Clinical Study of Merlin's DiVeRt - Vascular Reconstruction Device and Delivery System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Merlin MD Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VV0146
Record Dates: First submitted 2020-09-14; First posted 2020-10-19 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Intracranial Aneurysm, Wide Neck Aneurysm, Large Neck Aneurysm, Lesion
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DiVeRt treatment (Experimental): DiVeRt device to be used in the single arm
  Interventions: Device: DiVeRt

INTERVENTIONS:
Device: DiVeRt — DiVeRt - Vascular Reconstruction Device and Delivery System

SUMMARY:
The objective of the proposed investigation is to assess the safety and effectiveness of the Merlin's DiVeRt system for the treatment of intracranial lesions.

Merlin is a manufacturer of Flow- Diverters (FD) for Neurovascular applications. The technology is based on a microporous polymer membrane which is delivered to the site of lesion treatment using a metal stent scaffold. The first device in its FD family is the XCalibur Aneurysm Occlusion Device (AOD) system, which is delivered on a rapid-exchange balloon catheter which goes in a 6-Fr guide-catheter. The AOD is CE-marked and has been involved in the treatment of over 70 clinical lesion/aneurysm cases. The same technology is now being made available in a self-expandable stent platform delivered on a 0.028" microcatheter. Merlin has performed the required in-silico, in-vitro and in-vivo tests to be confident of the device performance and now intends to proceed to the human clinical-trials. DiVeRt (Interventional) is a non CE mark device. The device is under clinical trial phase. The competent authority submission for the study has been completed in Spain, Turkey and Hungary.

DETAILED DESCRIPTION:
The study will recruit patients with intracranial aneurysm (IA) or a lesion located in the anterior or posterior circulation. The analyses of the data from this safety and feasibility study will be descriptive.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent using the IRB/EC-approved consent form and agrees to comply with protocol requirements.
* Age 18-80 years.
* Subject has a target intracranial aneurysm (IA) or a lesion located in the anterior or posterior circulation.
* Subject has a target IA with a wide or large neck aneurysm or a lesion. The aneurysm type includes saccular, fusiform, dissecting or blister shapes.

Exclusion Criteria:

* Major surgery in the last 30 days.
* History of irreversible bleeding disorder and/or subject presents with signs of active bleeding.
* NIH Stroke Scale ( NIHSS) greater than or equal to 4
* Any known contraindication to treatment with flow diverters.
* Pregnant women.
* Participating in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of all serious adverse events assessed, clinically or angiographically | 3 months
  Serious Adverse events will be evaluated as device-related, procedure-related, or unrelated to the procedure or the device
Incidence of unsuccessful Divert placement | 3 months
  Incidence of unsuccessful Divert placement leading to, or with the potential of leading to, adverse events.
Aneurysm Occlusion Grading: MRRC scale | 3 months
  Evaluation of degree of aneurysm occlusion or degree of delayed opacification

SECONDARY OUTCOMES:
In-stent stenosis (DSA) | 6 months
  Evaluation of perforator vessel patency immediately post-implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Vall De Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No